CLINICAL TRIAL: NCT00268463
Title: A Phase III Clinical Trial Comparing Oxaliplatin, Capecitabine and Hepatic Arterial Infusion of Floxuridine to Oxaliplatin and Capecitabine in Patients With Resected or Ablated Liver Metastases From Colorectal Cancer
Brief Title: Oxaliplatin and Capecitabine With or Without an Hepatic Arterial Infusion With Floxuridine in Treating Patients Who Are Undergoing Surgery and/or Ablation for Liver Metastases Due to Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to low accrual.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP C-09; U10CA012027 (NIH)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Floxuridine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Capecitabine + Oxaliplatin (Active Comparator): Within 4-6 weeks after surgery and/or ablation, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: capecitabine; Drug: oxaliplatin
- Arm 2: Floxuridine + Oxaliplatin + Capecitabine (Experimental): Within 4-6 weeks after surgery and/or ablation, patients receive a continuous hepatic arterial infusion of floxuridine on days 1-14, oxaliplatin IV over 2 hours on day 22, and oral capecitabine twice daily on days 22-35. Treatment repeats every 42 days for 4 cycles in the absence of unacceptable toxicity. Beginning with cycle 5, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment with oxaliplatin and capecitabine repeats every 21 days for 4 cycles.
  Interventions: Drug: capecitabine; Drug: floxuridine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine — Oral capecitabine 850 mg/m2 twice daily on days 1-14 every 21 days for 8 cycles: Arm 1
  Oral capecitabine 850 mg/m2 twice daily on days 22-35 every 42 days for 4 cycles and then on days 1-14 every 21 days for 4 cycles: Arm 2
  Other Names: Xeloda
Drug: floxuridine — Continuous hepatic arterial infusion of floxuridine 0.2 mg/kg on days 1-14 every 42 days for 4 cycles
  Other Names: FUDR
  Arms: Arm 2: Floxuridine + Oxaliplatin + Capecitabine
Drug: oxaliplatin — Oxaliplatin 130 mg/m2 IV over 2 hours on day 1 every 21 days for 8 cycles: Arm 1
  Oxaliplatin 130 mg/m2 IV over 2 hours on day 22 every 42 days for 4 cycles and then on day 1 every 21 days for 4 cycles: Arm 2
  Other Names: Eloxatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, capecitabine, and floxuridine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Hepatic arterial infusion uses a catheter to carry tumor-killing substances, such as chemotherapy, directly into the liver. Giving chemotherapy in different ways may kill more tumor cells. It is not yet known whether giving oxaliplatin and capecitabine together with an hepatic arterial infusion with floxuridine is more effective than giving oxaliplatin and capecitabine alone in treating patients who are undergoing surgery and/or ablation for liver metastases due to colorectal cancer.

PURPOSE: This randomized phase III trial is studying oxaliplatin, capecitabine, and an hepatic arterial infusion with floxuridine to see how well they work compared to oxaliplatin and capecitabine in treating patients who are undergoing surgery and/or ablation for liver metastases due to colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free interval (PFI) in patients undergoing surgical resection and/or ablation for hepatic metastases from colorectal cancer treated with adjuvant therapy comprising oxaliplatin and capecitabine with vs without hepatic arterial infusion of floxuridine.

Secondary

* Compare overall survival and liver PFI between the two treatment groups.
* Assess toxicity in each of the treatment regimens.
* Compare self-reported symptoms between two treatment groups.
* Compare quality of life in each of the treatment regimens.

Tertiary

* Examine the prognostic worth, in terms of PFI, of specific molecular markers in hepatic metastases.

OUTLINE: This is a randomized study. Patients are stratified according to intended surgical technique (surgical resection alone vs cryoablation or radiofrequency ablation [RFA] alone vs combination of resection and ablation) and prior adjuvant chemotherapy regimen (chemotherapy with vs without oxaliplatin vs no chemotherapy). Patients are randomized to 1 of 2 treatment arms.

All patients undergo surgical resection and/or hepatic cryoablation or RFA to remove a maximum of 6 colorectal hepatic metastases. Patients randomized to arm II also undergo intra-arterial catheter and if applicable, pump placement.

* Arm 1 (oxaliplatin and capecitabine): Within 4-6 weeks after surgery and/or ablation, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
* Arm 2 (oxaliplatin, capecitabine, and hepatic arterial infusion of floxuridine): Within 4-6 weeks after surgery and/or ablation, patients receive a continuous hepatic arterial infusion of floxuridine on days 1-14, oxaliplatin IV over 2 hours on day 22, and oral capecitabine twice daily on days 22-35. Treatment repeats every 42 days for 4 courses in the absence of unacceptable toxicity. Beginning with course 5, patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment with oxaliplatin and capecitabine repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 4-6 weeks after surgery or ablation, approximately 18 weeks after beginning of chemotherapy, and 4-6 weeks after beginning the last cycle of chemotherapy.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* or cytologically confirmed colorectal adenocarcinoma

  * No other cellular type (e.g., sarcoma, lymphoma, or carcinoid) NOTE: *If the primary colorectal tumor and the hepatic lesions have been identified at the same time and it is not possible to biopsy the colorectal lesion, the patient will be eligible without histologic confirmation of the colorectal primary cancer as long as other radiographic studies or scans document the characteristics of a colorectal cancer
* Synchronous or metachronous metastatic disease confined to the liver

  * No more than 6 hepatic metastatic lesions that can potentially be resected or ablated
  * For patients presenting with synchronous lesion(s) in the colon and/or rectum, the primary tumors must, in the opinion of the investigator, appear to be completely resectable
* Must be able to undergo surgery and/or ablation within 28 days following randomization
* No evidence of extrahepatic metastases
* No prior colorectal metastases
* No recurrent colorectal cancer concurrent with hepatic metastases

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 5 years, excluding their colorectal cancer
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1
* No other malignancy within the past 5 years except carcinoma in situ of the cervix, melanoma in situ, basal cell or squamous cell skin cancer, or carcinoma of the colon or rectum
* Absolute granulocyte count ≥ 1,200/mm^3
* Platelet count ≥ 100,000/mm^3
* PT/international normalized ratio (INR) ≤ 1.5 unless patient is on therapeutic doses of anticoagulant medication
* Total bilirubin ≤ upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 ULN
* aspartate aminotransferase (AST) ≤ 2.5 times ULN
* Calculated creatinine clearance > 50 mL/min
* Not pregnant or lactating
* Negative pregnancy test
* Patients with child bearing potential must agree to use adequate contraception
* Able to swallow oral medication
* No preexisting chronic hepatic disease (e.g., chronic active hepatitis or cirrhosis)
* No grade 3 or 4 anorexia or nausea
* No vomiting ≥ grade 2
* No clinically significant peripheral neuropathy defined as ≥ grade 2 neurosensory or neuromotor toxicity
* No psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation

PRIOR CONCURRENT THERAPY:

* Prior adjuvant fluorouracil alone or in combination with levamisole, leucovorin calcium, irinotecan hydrochloride, or oxaliplatin allowed if these regimens were completed > 6 months ago
* No prior resection/ablation, hepatic arterial infusion therapy, or any systemic chemotherapy for metastatic disease

  * Prior excisional biopsy allowed
* No prior radiotherapy to the liver
* No concurrent bevacizumab in patients who have had pump/catheter placement receiving hepatic arterial infusion of floxuridine

  * Patients who meet specific situations outlined in the protocol and who have not had pump placement may receive bevacizumab at the physician's discretion
* No concurrent halogenated antiviral agents such as sorivudine or brivudine in patients receiving fluorouracil, floxuridine, or capecitabine
* No concurrent filgrastim (G-CSF), pegfilgrastim, or sargramostim (GM-CSF) as primary prophylaxis for neutropenia

  * Following neutropenic events, these drugs may be used at the physician's discretion during subsequent cycles
* No other concurrent cancer therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (31):
- United States (31):
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Center, Louisville, Kentucky
  - CCOP - Ochsner, New Orleans, Louisiana
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Capecitabine + Oxaliplatin: Oxaliplatin 130 mg/m2 IV over 2 hours on day 1 every 21 days for 8 cycles: Arm 1
  Oral capecitabine 850 mg/m2 twice daily on days 1-14 every 21 days for 8 cycles: Arm 1
- Arm 2: Floxuridine + Oxaliplatin + Capecitabine: Oxaliplatin 130 mg/m2 IV over 2 hours on day 22 every 42 days for 4 cycles and then on day 1 every 21 days for 4 cycles
  Oral capecitabine 850 mg/m2 twice daily on days 22-35 every 42 days for 4 cycles and then on days 1-14 every 21 days for 4 cycles
  Continuous hepatic arterial infusion of floxuridine 0.2 mg/kg on days 1-14 every 42 days for 4 cycles
Period: Overall Study
Arm/Group | Arm 1: Capecitabine + Oxaliplatin | Arm 2: Floxuridine + Oxaliplatin + Capecitabine
Started | 10 | 12
Completed | 0 | 0
Not Completed | 10 | 12
Not completed — study terminated due to low accrual | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Capecitabine + Oxaliplatin: Capecitabine + Oxaliplatin
- Floxuridine + Oxaliplatin + Capecitabine: Floxuridine + Oxaliplatin + Capecitabine
- Total: Total of all reporting groups
Arm/Group | Capecitabine + Oxaliplatin | Floxuridine + Oxaliplatin + Capecitabine | Total
Number analyzed (Participants) | 10 | 12 | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (10.4) | 59 (9.4) | 59 (9.7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 3 | 4 | 7
  Male | 7 | 7 | 14
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Interval (PFI)
Description: Time to first recurrence of colon cancer at any site
Time Frame: Time from randomization through year 5
Arm/Group | Arm 1: Capecitabine + Oxaliplatin | Arm 2: Floxuridine + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Liver PFI as Measured by Time to Hepatic Progression.
Time Frame: Time from randomization through year 5
Reporting Status: Not Posted

3. Secondary Outcome: Survival as Measured by Time to Death From Any Cause.
Time Frame: Time from randomization through year 5
Reporting Status: Not Posted

4. Secondary Outcome: Scales Specific to Social/Family, Emotional, and Functional Well-being, Perceived Convenience of Care, and Self-reported Symptoms
Time Frame: Prior to randomization, 4-6 weeks after surgery, 18 weeks after starting chemotherapy and after completion of chemotherapy
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life as Measured by the Functional Assessment of Cancer Therapy Trial Outcome Index at Baseline, at 4-6 Weeks Following Surgery (Before Initiation of Chemotherapy), and Periodically During Study
Time Frame: Prior to randomization, 4-6 weeks after surgery, 18 weeks after the start of chemotherapy and after completion of chemotherapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Arm/Group | Capecitabine + Oxaliplatin | Floxuridine + Oxaliplatin + Capecitabine
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 6/8 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Oxaliplatin (N=8) | Floxuridine + Oxaliplatin + Capecitabine (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Fatigue (General disorders) | 0 | 2
Fever (General disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Neutrophil count decreased (Investigations) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less